CLINICAL TRIAL: NCT04147026
Title: PRediction mEdical DevIce for Rheumatoid Arthritis: Scale-up of Unique Predictive Online Platform Highly Improving the Quality of Life of Rheumatoid Arthritis' Patient by Personalised and Efficient Biotherapies Prescription
Brief Title: Prediction Medical Device for Rheumatoid Arthritis (PREDIRA)
Acronym: PREDIRA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Benjamin Fernandez Gutierrez, Principal Investigator, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EUR.PREDIRA
Record Dates: First submitted 2019-10-25; First posted 2019-10-31 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Arthritis, Rheumatoid
Keywords: Biological therapy; Predictive software; Quality of life
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: The study is a prospective, phase III, controlled, multicenter, and randomized in 2 parallel groups, single-blind (patient) with binded outcome assessment clinical trial.
  * Intervention arm: Prescription of biotherapy (rituximab, adalimumab, abatacept) using SinnoTest® software
  * Control arm: Prescription of biotherapy without the SinnoTest® software which corresponds to current practice (all biotherapies).
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient will not know if his bDMARD treatment was prescribed with or without the help of SinnoTest® software
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SinnoTest® software (Experimental): SinnoTest® is a therapeutic guidance device for patients suffering from rheumatoid arthritis. Prescription of an original or biosimilar biotherapy (rituximab, adalimumab, abatacept) is possible.
  Interventions: Device: SinnoTest®
- Current practice (Active Comparator): Prescription of biotherapy without the SinnoTest® software which corresponds to current practice (all biotherapies).
  Interventions: Other: Biotherapy prescription without SinnoTest® software

INTERVENTIONS:
Device: SinnoTest® — The selection of the biotherapy is carried out based on the recommendations of SinnoTest®. This test categorizes the bDMARDs based on the probability of response. It will allow to prescribe both original molecules, as well as biosimilars, in an equivalent way.
  In the SinnoTest® arm, the investigator prescribes the treatment defined as the most effective by SinnoTest®, except in case of contraindication. If contraindicated, the investigator prescribes the second-choice treatment (if any) of SinnoTest® in terms of efficacy.
  Arms: SinnoTest® software
Other: Biotherapy prescription without SinnoTest® software — The rheumatologist will use the current guidelines of rheumatoid arthritis to choose the more adapted biotherapy treatment to the patient
  Arms: Current practice

SUMMARY:
Rheumatoid arthritis (RA) is one of the leading chronic inflammatory rheumatism, with a prevalence of about 0.4% of the population.

First-line therapy with synthetic disease modifying anti-rheumatic drugs (including methotrexate) is insufficiently effective in 40% of cases. These patients are then treated with biotherapies. The use of these bio-drugs increases each year, becoming a public health issue and a considerable economic burden. Besides, their growth is just beginning, as they are among the major purveyors of pharmacy innovations.

There are about ten bio-drugs currently on the market for rheumatoid arthritis with an average annual treatment cost of 8 to 12 K € per patient. This cost is 20 times higher than that of synthetic disease modifying anti-rheumatic drugs. However, among patients treated with biotherapies, clinical practice shows that about one-third will not respond to the selected drug. In the case of non-response, practitioners currently have no choice but to perform an empirical rotation between the different treatments, because no tool capable of predicting the response or non-response to these molecules is currently available.

The study is a prospective, phase III, controlled, multicenter, and randomized, single-blind (patient) clinical trial.

* Intervention arm: Prescription of biotherapy (rituximab, adalimumab, abatacept) using SinnoTest® software
* Control arm: Prescription of biotherapy without the SinnoTest® software which corresponds to current practice (all biotherapies).

In addition, a sub study will be carried out within this trial to analyse the proteomic profile of the patients included and their modification throughout the study.

To study the clinical and pharmacoeconomic impact after 6 months of the use of the SinnoTest® predictive tool in patients with rheumatoid arthritis who have failed to a first anti-TNF biologic agent compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old and under 70 years old,
* Patients with RA, defined according to the ACR / EULAR 2010 or ACR 1987 criteria,
* Patients failing a first anti-TNF, defined as:
* Ineffectiveness (which is defined as a DAS28-ESR ≥3.2 and an inadequate response to iTNF according to the usual rheumatologist, which generally includes one or more of the following conditions: persistent swollen and tender joints, persistence of disease activity according to the overall evaluation of the patient, high levels of acute phase reactants and/or dependence of analgesics, nonsteroidal anti-inflammatory drugs or corticosteroids); or
* Toxicity(defined as the appearance of any adverse event that the patient's rheumatologist relates to the medication and requires discontinuation),
* Effective contraception for patients of childbearing potential (oral contraceptive, intrauterine device, implant, spermicide, surgical sterilization or abstinence),
* Patients able to read and understand the modalities of the protocol,
* Patients who have dated and signed the informed consent form of the trial,
* Stability of treatments (no change) between the selection visit and the inclusion visit (M0).

Exclusion Criteria:

* Patients with a contraindication to any bDMARD or methotrexate,
* Patients included in another therapeutic evaluation study during this trial,
* Surgical intervention programmed during the trial,
* Patients with difficulties in understanding the Spanish language,
* Patients cannot be followed up 6 months,
* Psychosocial instability incompatible with regular monitoring (homelessness, addictive behaviour, antecedent of psychiatric pathology or any other comorbidity that would make it impossible for free and informed consent or limit adherence to the protocol),
* Breastfeeding and/or pregnancy. Although there are bDMARD that can be used in pregnancy, since SinnoTest can recommend one that discourages this condition, it is decided to exclude the inclusion of pregnant women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Incremental Cost Utility ratio at 6 months | 6 months
  This outcome will be calculated as the average differential cost per patient between both study arms (mean costs of the Sinnotest® Arm - mean costs of the Control Arm) divided by the diference in effectiveness between both study arms measured in the number of years of life weighted by the quality of life (QALY: quality-adjusted life year) generated by each of the strategies (mean QALY of the Sinnotest® Arm - mean QALY of the Control Arm).
  QALY will be measured using the EuroQol-5D. Cost will be considered from a Societal perspective, including both direct and indirect costs The ratio will be expressed in cost (2019 Euros) per QALY earned, which represents the additional cost that will have to be spent to earn a healthy year of life

SECONDARY OUTCOMES:
Budget impact analysis at 6 and 12 months | 12 months
  A budget impact analysis will be carried out if the innovation is deemed efficient.
  This budget impact analysis will describe the resources consumed and the expenses generated by each scenario, a scenario with the use of SinnoTest® and a scenario without SinnoTest®.
Software's predictive model performance | 6 months
  Sensitivity, Especificity, positve and negative preddicted values of the predictive models using the biomarkers will be assessed on the new clinical data from the 6-month trial.
Description of the variation of the proteomic profile between M0 (biotherapy start date) and M6 (6 months visit) | Inclusion and 6 months
  Based on shotgun and semiquantitative proteomics, the diferences between the proteomic profile at baseline and at M6 will be analyzed

OTHER OUTCOMES:
Incremental Cost Effectiveness ratio at 6 months | 6 months
  This outcome will be calculated as the average differential cost per patient between both study arms (mean costs of the Sinnotest® Arm - mean costs of the Control Arm) divided by the diference in effectiveness between both study arms measured as the percentage of patients achieving a good clinical response in each study arm (% in the Sinnotest® Arm - % in the Control Arm).
  Good clinical response will be measured using the EULAR criteria of Good clinical response Cost will be considered from a Societal perspective, including both direct and indirect costs The ratio will be expressed in cost (2019 Euros) per increase in 1% of subjects achieving a Good Clinical Response, which represents the additional cost that will have to be spent to earn a healthy year of life
  rates of treatment-response patients associated respectively with the usual strategy without SinnoTest® and with the strategy with SinnoTest®

CONTACTS AND LOCATIONS:
Overall Officials: Benjamín Fernández-Gutiérrez, MD, PhD, Principal Investigator — Hospital San Carlos, Madrid
Locations (5):
- Spain (5):
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de La Paz, Madrid

REFERENCES:
- [Background] Nguyen MVC, Baillet A, Romand X, Trocme C, Courtier A, Marotte H, Thomas T, Soubrier M, Miossec P, Tebib J, Grange L, Toussaint B, Lequerre T, Vittecoq O, Gaudin P. Prealbumin, platelet factor 4 and S100A12 combination at baseline predicts good response to TNF alpha inhibitors in rheumatoid arthritis. Joint Bone Spine. 2019 Mar;86(2):195-201. doi: 10.1016/j.jbspin.2018.05.006. Epub 2018 Jun 6. PMID 29885551
- [Background] Nguyen MVC, Adrait A, Baillet A, Trocme C, Gottenberg JE, Gaudin P. Identification of cartilage oligomeric matrix protein as biomarker predicting abatacept response in rheumatoid arthritis patients with insufficient response to a first anti-TNFalpha treatment. Joint Bone Spine. 2019 May;86(3):401-403. doi: 10.1016/j.jbspin.2018.09.005. Epub 2018 Sep 19. No abstract available. PMID 30243783
- [Background] Baillet A, Trocme C, Romand X, Nguyen CMV, Courtier A, Toussaint B, Gaudin P, Epaulard O. Calprotectin discriminates septic arthritis from pseudogout and rheumatoid arthritis. Rheumatology (Oxford). 2019 Sep 1;58(9):1644-1648. doi: 10.1093/rheumatology/kez098. PMID 30919904
- [Background] Baillet A, Trocme C, Berthier S, Arlotto M, Grange L, Chenau J, Quetant S, Seve M, Berger F, Juvin R, Morel F, Gaudin P. Synovial fluid proteomic fingerprint: S100A8, S100A9 and S100A12 proteins discriminate rheumatoid arthritis from other inflammatory joint diseases. Rheumatology (Oxford). 2010 Apr;49(4):671-82. doi: 10.1093/rheumatology/kep452. Epub 2010 Jan 25. PMID 20100792
- [Background] Trocme C, Marotte H, Baillet A, Pallot-Prades B, Garin J, Grange L, Miossec P, Tebib J, Berger F, Nissen MJ, Juvin R, Morel F, Gaudin P. Apolipoprotein A-I and platelet factor 4 are biomarkers for infliximab response in rheumatoid arthritis. Ann Rheum Dis. 2009 Aug;68(8):1328-33. doi: 10.1136/ard.2008.093153. Epub 2008 Jul 29. PMID 18664547
- [Derived] Freites-Nunez D, Baillet A, Rodriguez-Rodriguez L, Nguyen MVC, Gonzalez I, Pablos JL, Balsa A, Vazquez M, Gaudin P, Fernandez-Gutierrez B. Efficacy, safety and cost-effectiveness of a web-based platform delivering the results of a biomarker-based predictive model of biotherapy response for rheumatoid arthritis patients: a protocol for a randomized multicenter single-blind active controlled clinical trial (PREDIRA). Trials. 2020 Aug 31;21(1):755. doi: 10.1186/s13063-020-04683-7. PMID 32867830